CLINICAL TRIAL: NCT00003796
Title: Phase II Study of MGI-114 in Patients With Metastatic Breast Cancer
Brief Title: Irofulven in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066939; UTHSC-IDD-98-23; SACI-IDD-98-23; NCI-T98-0060
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2003-03

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — irofulven

ARMS (1):
- Arm I (Experimental): Patients receive irofulven IV over 30 minutes on days 1 and 15. Treatment continues every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: irofulven

INTERVENTIONS:
Drug: irofulven

SUMMARY:
Phase II trial to study the effectiveness of irofulven in treating patients who have metastatic breast cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Evaluate the response rate and time to treatment failure in patients with refractory metastatic adenocarcinoma of the breast treated with irofulven.

II. Assess the qualitative and quantitative toxic effects of this drug in these patients.

III. Determine the population pharmacokinetics and the pharmacokinetics-pharmacodynamic relationships of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive irofulven IV over 30 minutes on days 1 and 15. Treatment continues every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic adenocarcinoma of the breast
* Measurable disease outside previously irradiated area or occurred/progressed after completion of radiotherapy
* Must have received 1 or 2 prior chemotherapy regimens for metastatic disease

  * More than 3 prior regimens allowed
* No active brain metastases or meningeal breast cancer involvement

PATIENT CHARACTERISTICS:

Sex:

* Male or female

Performance status:

* SWOG 0-2

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT or SGPT no greater than 3 times ULN (5 times ULN for liver metastases)

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No history of myocardial infarction or unstable angina within the past 6 months
* No uncontrolled congestive heart failure

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Prior diagnosis of cancer allowed (must be off cancer therapy and have no evidence of disease)
* No history of retinopathy and/or macular degeneration

PRIOR CONCURRENT THERAPY:

Chemotherapy:

* No prior irofulven

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 1999-05; Primary Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hammond, MD, Study Chair — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States